CLINICAL TRIAL: NCT00614822
Title: A Phase II Trial of Carboplatin, Bevacizumab and Pemetrexed in Advanced Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Bevacizumab and Pemetrexed in Advanced Non Small Cell Lung Cancer
Acronym: H3E-US-X072
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24091; Eli Lilly H3E-US-X072 (Other Grant/Funding Number: Eli Lilly)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm for study (Other): Carboplatin, Pemetrexed and Bevacizumab are given day 1 every 3 weeks for 6 cycles and will be continued if patient tolerates treatments and has stable disease. The Bevacizumab will be continued every 3 weeks for 1 year if the patient tolerates treatment and has stable disease.
  Interventions: Drug: Carboplatin, Pemetrexed and Bevacizumab

INTERVENTIONS:
Drug: Carboplatin, Pemetrexed and Bevacizumab — Carboplatin AUC 5 IV day 1 over 30-60 minutes Pemetrexed 500 mg/M2 IV day 1 over 10 minutes Bevacizumab 15 mg /kg IV day over 90 minutes dose 1, 60 minutes dose 2, 30 minutes subsequent doses. Repeat every 3 weeks for total of 6 cycles
  Other Names: Paraplatin; Alimta; Avastin

SUMMARY:
The purpose of this study is to look for an improvement in progression free survival with the combination of bevacizumab, carboplatin and pemetrexed in patients with newly diagnosed advanced/metastatic non small cell lung cancer. Overall survival and safety will also be assessed.

DETAILED DESCRIPTION:
Carboplatin: AUC 5 IV over 30-60 minutes on day 1 Pemetrexed: 500mg/M2 IV over 10 minutes on day 1 Bevacizumab: 15mg/kg IV over 90 minutes on day 1 (if rate is tolerated the 2nd dose may be decreased to 60 minutes and subsequent doses to 30 minutes This regimen will be administered every 6 weeks for up to a maximum of 6 cycles if the patient tolerates the treatment and has stable disease. Bevacizumab will be continues if tolerated for up to 1 year at every 3 week intervals.

Folic acid 1mg by mouth daily, Vitamin B12 1000 ug IM every 9 weeks and Dexamethasone 4mg by mouth twice a day and and antiemetic may be prescribed by the physician investigator to help reduce side effects associated with the Pemetrexed. The Folic acid and Vitamin B12 will continue until 3 weeks after the end of treatment.

Physical exams, vital signs and blood work will be done prior to each chemotherapy cycle. A urine dipstick to check for protein in the urine will be done prior to the first treatment and before cycles 3 and 5. A CAT scan of the chest will be done pretreatment, prior to cycles 3 and 5 and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage NSCLC (IIIB with malignant pleural effusion; T4 [on basis on satellite lesion] N2, 3; or stage IV) excluding squamous cell histology, with measurable or evaluable disease.
* Prior chemotherapy therapy for early stage disease with one regimen is acceptable if it was completed at least 6 months prior to study entry.
* Palliative radiotherapy to painful bony metastases will be permitted prior to study entry if completed prior to initiation of study treatment, and there are no residual sequelae of therapy such as bone marrow suppression.
* Life expectancy of at least 3 months.
* ECOG Performance status 0-1.
* Age 18 or higher.
* Willingness to use appropriate contraception to avoid pregnancy during the study (female patient or female partner of a male patient)
* Patients must have normal organ and marrow function as defined below:

leukocytes greater than or equal to3,000/µl ANC greater than or equal to 1,500/µl platelets greater than or equal to 100,000/µl total bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal creatinine within normal institutional limits OR creatinine clearance ≥ 45 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

* Ability to sign informed consent
* Ability to take folic acid, Vitamin B12 and dexamethasone as per protocol
* Ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Alimta.

Exclusion criteria

Patients meeting any of the following criteria are ineligible for study entry:

* Prior cytotoxic treatment for advanced NSCLC. One prior regimen (up to 4 cycles) of neoadjuvant or adjuvant therapy for early stage disease will be allowed if completed at least 6 months prior to study entry.
* Prior definitive chest irradiation (radiation of rib or spine mets permitted)
* Known brain metastases (unless previously resected and radiated)
* Prior treatment with bevacizumab or pemetrexed
* History of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to bevacizumab or carboplatin
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in any other experimental drug study.
* Concomitant chemotherapy, radiotherapy or investigational agents.
* Evidence of bleeding diathesis or coagulopathy.
* Use of anti-coagulant agents warfarin (1mg, by mouth, daily for port maintenance permitted), heparin (ASA, NSAID permitted).
* Pregnant (positive pregnancy test) or lactating women.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0.
* Urine protein creatinine ratio 1.0 at screening. -History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 6 months prior to Day 0.
* Serious, non-healing wound, ulcer, or bone fracture.
* Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, or with significant cavitation as assessed by treating investigator in consultation with an attending radiologist. -Recent history of hemoptysis (bright red blood of 1/2 teaspoon or more)- within one month of study entry
* Significant co-morbidities including:

Blood pressure of 150/100 mmHg Unstable angina New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix B) History of myocardial infarction within 6 months History of stroke within 6 months Clinically significant peripheral vascular disease

* Psychiatric illness/social situations that would limit compliance with study requirements.
* Another active malignancy except for non-melanoma skin cancers.
* Clinically significant pleural, pericardial, and/or peritoneal effusions unless drained or controlled prior to study entry.
* Undrainable, clinically relevant effusions and presence of third space fluid which cannot be controlled by drainage.
* Hepatic impairment as evidenced by Bilirubin greater than 1.5 times the upper limit of normal Transaminases greater than 3.0 times limit of normal (ULN), except in presence of known hepatic metastasis, wherein may be up to 5 times ULN
* Any CTCAE Version 3.0 Grade 3 or 4 non hematologic toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Guarino, MD, Principal Investigator — Christiana Care Health Services

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2007 and March 2012, 50 patients were enrolled in the phase II trial of carboplatin, pemetrexed and bevacizumab. Patients were enrolled over a 24month period.
Pre-assignment Details: Carboplatin, Penetrexed and Bevacizumab in Advanced Non-Squamous Non-Small Cell Lung Cancer
Period: Overall Study
Arm/Group | One Arm for Study
Started | 50
Completed | 47
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- Carboplatin, Bevacicumab, Premetrexed: Patients (age >18yo) were from 2007 to 2012.. Measurable disease Evaluable disease Stage IV Palliative RT NO brain metastases
Arm/Group | Carboplatin, Bevacicumab, Premetrexed
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  SEX: Female | 24
  SEX: Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance [Count of Participants; unit: Participants] — ECOG Performance Status Scale are measurements of a patient's status. ECOG 0 = Fully active, able to carry on all pre-disease performance without restriction ECOG 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG Performance Staus Scale 0 | 6
    ECOG Performance Stsus Scale =1 | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year").
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year").
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Carboplatin, Bevacicumab, Premetrexed: Patients (age >18yo) were from 2007 to 2012.. 51 patients with nonsquamous stage IV disease were enrolled over 24 months and followed. The meadian follow up was 49 weeks. Of the 51 patient enrolled, 1 patient was with drawn due to ineligibility. Three other patients were not evaluated for response due to adverse reactions.
Arm/Group | Carboplatin, Bevacicumab, Premetrexed
Number analyzed (Participants) | 47
weeks | 28 [0 to 132.4]

2. Primary Outcome: Overall Survival
Description: Overal survival was defined as time between the date of treatment assignment and the date of death
Time Frame: as for outcome 1
Population: Nonsquamous stage IV disease, Male, Female,>18 years of age, white, african american,with ECOG of 0 or 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | One Arm for Study
Number analyzed (Participants) | 47
weeks | 49 [0 to 62.7]

3. Secondary Outcome: Number of Participants With Complete and Partial Tumor Responses
Description: A complete response (CR),was disappearance of all target lesions on CT scan and absence of appearance of any new lesion was required. Partial response (PR) was assessed by at least a 30% decrease in the sum of the longest diameter (LD) of target lesions without appearance of any new lesions. Progressive disease (PD) was defined as at least a 20% increase in the sum of the LD of target lesions or the appearance of one or more new lesions. Patients were assessed to have stable disease if neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD, without appearance of new lesions. Patients who received one or more cycles were evaluable for response.
Time Frame: Patients were enrolled over a 24 month period for treatment visits. After end of treatment visits, subjects were seen or contacted every 3 months for survival data. Median follow up was 49 weeks (6 weeks to death.
Population: Number of Participants with Complete and Partial Tumor Responses
Measure: Count of Participants; unit: Participants
Arm/Group | One Arm for Study
Number analyzed (Participants) | 47
Participants
  Complete Response | 1
  Partial Response | 27

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Measured by adverse events such as grade 4 toxicities, hospitalizations for toxicities, fever and neutropenia events, and clinically significant bleeding/thrombotic events.
Time Frame: Subjects were seen or contacted every 3 months with medain follow up of 49 weeks.
Population: four patients discontinued treatment because of treatment related adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | One Arm for Study
Number analyzed (Participants) | 47
Participants
  Thrombocytopenia | 1
  Respiratory distress | 1
  Grade 3 diarrhea | 1
  fatigue | 1

ADVERSE EVENTS:
Arm/Group | One Arm for Study
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Arm for Study (N=50)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
grade 3 Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Arm for Study (N=50)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
include the absence of randomization, lack of independent radiology review and small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No